CLINICAL TRIAL: NCT05536843
Title: Circulating Cell-Free Tumor Tissue Modified Viral (TTMV)-HPV DNA As A Biomarker For Early Cancer Detection Among Human Subjects With HPV-Induced Dysplasia In Female Genital [Uterine Cervix, Vaginal and Vulvar] Organs: A Clinical, Translational and Biomarker-Based Cancer Screening Study
Brief Title: Clinical, Translational and Biomarker-Based Female Genital HPV Induced Dysplasia and Cancer Screening Study Using Cf-HPV-DNA Blood Tests
Acronym: TTMV HPV DNA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMississippiRadOnc
Record Dates: First submitted 2022-09-07; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Cervical Dysplasia, Uterine; Vaginal Dysplasia; Vulvar Dysplasia
Keywords: HPV; Dysplasia; Liquid Biopsy; Screening; Female Genital Cancer
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Blood collection from the subject vein by UMMC's trained professionals of about four table spoons of blood like for any other blood test.
  2. The samples collected will be frozen and stored to be utilized in the future for research studies. These samples will be labeled using a key code instead of the subject name, and no one using these samples for future research will know your name.
  3. Touch Preparation from the subject genital lesion being taken by our clinical care providers.
  Our research personnel will collect relevant information from your electronic medical records. The samples collected in this study could be used for genetic research studies. However, these results will not be added to your medical records. The samples collected in this study could be used to develop new treatments, drugs, or for other commercial purposes/third party company
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Uterine cervical dysplasia and other female genital dysplasia continue to be significant health problems despite Cervical Screening Programs and HPV vaccinations being available. These female genital dysplasia [FGD] induced by HPV infections affect disadvantaged women in the US and globally more than others: minorities like African Americans [AA], rural populations, lower socioeconomic strata of the society and less educated in the US and lower / middle income countries. The reasons are: lack of access to screening and vaccines, lack of infrastructure, fear and shame of getting a pelvic examination and pap's smear and inability to go to the health centers that provide these cares. A simple blood test that can diagnose FGD can help make many of those hurdles go away. This proposal is to utilize the emergence of 'liquid biopsy' concepts using genomic/precision medicine advances of the past decade to have such a blood test to be made available. Collaborating with Naveris, Inc,® the clinical study will use their NavDx® blood test. This is a test for circulating cell-free tumor tissue modified viral (TTMV®)-HPV DNA. TTMV-HPV DNA is a clinically proven and analytically validated highly sensitive and specific biomarker for the identification of post-treatment recurrent and residual Human Papillomavirus (HPV)-driven squamous cell oropharyngeal carcinoma (OPSCC)1,2. Data is accruing for other major HPV-driven cancers including anal cancer and uterine cervical cancer with clinical utility appear similarly promising3. TTMV-HPV DNA is a distinct biomarker for HPV-driven malignancy and can distinguish between HPV-driven malignancy and acute and or chronic HPV infection. In this study, taking advantage of a robust Cervical Dysplasia Clinic in existence at UMMC and a team of multidisciplinary experts focused on this project, the blood levels of TTMV-HPV DNA will be determined through a fully informed IRB approved clinical trial process to correlate with the grades of dysplasia, any increasing values correlating with worsening grade/malignant transformation and other variables. This pilot study is the first of this type of biomarker-based 'screening' study, and if successful, will lead to a more efficient and convenient way to diagnose HPV-induced that will be cost effective and will need minimal infrastructure. Such a test will make remarkable beneficial differences in early diagnosis, early screening compliance, early interventions as well as improving outcomes in FGD patients worldwide. With the available infrastructure and expert team, this project can be successfully completed in a relatively short time.

DETAILED DESCRIPTION:
Hypothesis:

1. The HPV induced dysplasia in cervical and vaginal tissues can lead to a detectable level of TTMV-HPV-DNA in the blood.
2. Those levels will increase when there is progression of the dysplasia from lower grade to a higher grade.
3. The blood levels of TTMV-HPV-DNA can distinguish lower versus higher grades of HPV induced dysplasia.
4. Serial measurements of TTMV-HPV-DNA in the blood can help diagnose progression of dysplasia to a higher grade earlier and in a more efficient and convenient way. This will help improved compliance with screening, early diagnosis, early interventions, and better clinical outcomes.
5. TTMV-HPV-DNA detection is also likely possible with touch preparations on the lesions, thus leading to easier diagnosis of such lesions.

Specific Aims:

1. To collect blood and touch-preparation samples from the dysplasia lesions among patients with HPV induced dysplasia in cervical and vaginal tissues in human subjects with such lesions in a phase I/II clinical trial setting.
2. Measure TTMV-HPV-DNA in those samples.
3. Correlate the detectable levels of TTMV-HPV-DNA with demographics, grades of dysplasia, progression in the grades with serial measurements and HIV status and correlate with biopsy results in terms of progression in PIN grades and malignant transformation.
4. Design future studies from these findings to enable early detection of potential progression to malignancy so that early curative interventions can be instituted.

Objectives:

1. To develop an innovative and pilot clinical trial in HPV related female genital dysplasia that integrates basic science, public health, clinical and translational cutting-edge knowledge and information using 'liquid biopsy' concepts to help prevent progression to malignancy.
2. To collect and analyze data in a prospective manner among a diverse population in terms of ethnic, racial, and socioeconomic variations that could help improve screening acceptance in the most vulnerable women at risk for female genital cancer.
3. To serve as a model for middle and low-income countries as well as resource-scarce, rural and disparity-affected populations in high-income countries in developing a blood-specimen based HPV-related early diagnosis screening tool.

ELIGIBILITY:
Inclusion Criteria:

* Adult women with female genital dysplasia
* Non pregnant women
* No prisoners
* age in between 18 years and 100 years
* Competent to give informed consent

Exclusion Criteria:

* Pregnant women
* Female below 18 years
* Prisoners

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult women with female genital dysplasia; Non pregnant women; No prisoners; Competent to give informed consent
Study Population: Adult non-pregnant women diagnosed with female genital dysplasia at the University of Mississippi Medical Center
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
CORRELATION BETWEEN BLOOD BASED 'LIQUID BIOPSY' BIOMARKER TO TISSUE DIAGNOSIS | 1 year
  Correlate the detectable levels of TTMV-HPV-DNA with demographics, grades of dysplasia, progression in the grades with serial measurements and HIV status and correlate with biopsy results in terms of progression in PIN grades and malignant transformation.
  Given the pilot nature of the proposed study, extensive use of exploratory data analysis will be done. For any analysis of time-to-event data,Kaplan-Meier analyses paired with two-sided log-rank tests will be used. For any necessary modeling, a generalized linear model framework will be employed with appropriate family and link functions, depending on the outcome. Should independence fail between the sampling units (repeated measures, etc.), this will be extended to generalized linear mixed models with random intercepts. All linearity assumptions will be checked and modifications to modeling strategies will be undertaken where necessary."